CLINICAL TRIAL: NCT05612061
Title: Randomized Controlled Trial of Indigenous Recovery Planning for American Indians
Brief Title: Indigenous Recovery Planning for American Indians
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01DA053791-02 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Wait-list control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Receives Indigenous Recovery Planning (IRP) intervention, which includes 6 weekly group intervention sessions lasting about 2 hours each.
  Interventions: Behavioral: Indigenous Recovery Planning
- Waitlist Control Group (No Intervention): Participants in the waitlist control group do not receive the intervention until after treatment group completes the intervention. Outcomes will be compared between the 2 study arms at baseline and at follow-up, at which point the treatment group will have completed the intervention and the waitlist control group will have not yet been exposed to the intervention, thereby serving as the control group.

INTERVENTIONS:
Behavioral: Indigenous Recovery Planning — The Indigenous Recovery Planning (IRP) intervention consists of a 6-week group-based intervention. Each of the 6 weekly sessions is delivered by a community member facilitator. Facilitators lead the group through a series of culturally adapted relapse prevention exercises designed to change their substance use.
  Focus areas for the 6 sessions are: 1) introduction and goal setting; 2) relapse and recovery; 3) craving, mindfulness, and self-compassion; 4) coping with trauma and stress; 5) enlisting social support for recovery; 6) envisioning and planning for the future.
  Arms: Treatment Group

SUMMARY:
This research project uses a Community-Based Participatory Research (CBPR) framework to test the efficacy of a culturally adapted relapse prevention intervention developed collaboratively by community partners from the Fort Peck Indian Reservation in northeastern Montana and research partners from Montana State University. The Indigenous Recovery Planning intervention employs trained Fort Peck community members to deliver manualized intervention content to American Indian adults with substance use disorder (SUD). By increasing access to culturally responsive evidence-based treatment, this research aims to decrease SUD-related health disparities and improve public health outcomes for underserved Native communities locally and nationally.

ELIGIBILITY:
Inclusion Criteria:

* American Indian, 18 years of age or older, living on the Fort Peck reservation, meeting diagnostic criteria for Substance Use Disorder, wanting treatment/help with recovery.

Exclusion Criteria:

* Not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percent days absent | At Time 1, we will assess alcohol and drug use in the 90 days prior to assessment, and each subsequent assessment will measure use in the time since the previous one (approximately 6 weeks).
  Percent days absent will be measured using the Timeline Followback (TLFB), a widely used calendar-based recall instrument shown to yield valid and reliable estimates of substance use behavior. Additional analyses will be conducted with other variables derived from TLFB data, including number of drinks per drinking day, percent heavy drinking days, and percent drug use days.

SECONDARY OUTCOMES:
Number of substance-related consequences experienced within the past 6 weeks | Measured at baseline and each 6 week follow-up assessment time point (time 1-time 5)
  Measured by the Drinker Inventory of Consequences, modified for alcohol and drug use

OTHER OUTCOMES:
Quality of life score | Measured at baseline and each 6 week follow-up assessment time point (time 1-time 5)
  Measured by the World Health Organization Brief Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Monica Skewes, PhD, Principal Investigator — Montana State University
Locations (1):
- Fort Peck Community College, Poplar, Montana, United States

IPD SHARING:
Plan to Share IPD: No
The data belong to the tribal community; data may be shared upon request to the tribe.